CLINICAL TRIAL: NCT04121039
Title: A Randomized,Parallel Controlled,Multicentre,Phase II Study of Apatinib Plus POF (Paclitaxel Plus Oxaliplatin Plus 5-fluorouracil Plus Leucovorin) Versus POF in Patients With Advanced/Metastatic Bastric Cancer
Brief Title: Study of the Apatinib Combine With POF Versus POF in Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF016
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Gastric Adenocarcinoma; Advanced Cancer
MeSH Terms: interventions — apatinib; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apatinib plus POF (Experimental): Participants will receive apatinib in combination with POF,total 9-12 cycles.Then receive apatinib plus S-1 until pre-defined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Apatinib
- POF (Active Comparator): Participants will receive POF,total 9-12 cycles.Then receive S-1 until pre-defined study end, disease progression, unacceptable toxicity, withdrawal of consent or death, whichever occurs first.
  Interventions: Drug: Apatinib; Drug: POF

INTERVENTIONS:
Drug: Apatinib — Apatinib (500 mg qd p.o.) until disease progression or intolerable toxicity or refused by the patients.
  Other Names: Study drug
Drug: POF — The POF regimen consisted of a 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.
  Arms: POF

SUMMARY:
This study is a randomized, parallel control, multicenter,phase II study, comparing the efficacy and safety of apatinib plus POF(paclitaxel plus oxaliplatin plus 5-fluorouracil plus leucovorin) versus POF, in the first-line treatment for patients with advanced/metastatic gastric cancer.

DETAILED DESCRIPTION:
This is a randomized, two-arm, open-label, multicenter phase II trial. Our primary purpose is to compare that PFS rate at 6-month of patients with apatinib plus POF and POF for advanced/metastatic gastric cancer.

Eligible patients will randomized to a ratio of 1:1 to apatinib+POF (experimental group) or POF (control group). Stratification factors were 1) gender (male;female);2) previous surgical history (yes;no);3) metastatic sites (measurable; Immeasurable).

In treatment period, patients will be administrated POF, with or without apatinib, every 14 days for 1 cycle, total 9-12 cycles.After the above treatment finished,parients will received with S-1,with or without apatinib,every 21days for 1 cycle,until disease progression, toxicity intolerance, withdrawal of informed consent, patients judged must be terminated study termination.

The imaging evaluation was performed according to the RECIST 1.1 criteria every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced unresectable, histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction.

No previous treatment with chemotherapy or radiation therapy. Ability to take medications orally. With measurable lesions. Patients must have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.

Without serious system dysfunction and could tolerate chemotherapy. With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥100g/L (without blood transfusion during 14 days); a leucopenia count of ≥4.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.

Life expectancy ≥3 months. With normal electrocardiogram results and no history of congestive heart failure.

Without bleeding and thrombosis disease. With normal coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT) and INR, each ≤ 1.5 x ULN.

Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.

With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

* Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.

Patients with brain or central nervous system metastases, including leptomeningeal disease.

Pregnant (positive pregnancy test) or breast feeding. Serious, non-healing wound, ulcer, or bone fracture. Significant cardiac disease as defined as: unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months Evidence of bleeding diathesis or coagulopathy.

History of a stroke or CVA within 6 months. Clinically significant peripheral vascular disease. Inability to comply with study and/or follow-up procedures. Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Rate at 6-month | Up to approximately 6 months
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.PFS rate at 6-month defined from randomization to 6 month,the cases of patients documented no PD or death or not receive other anti-tumor treatment in percentage of evaluable patients

SECONDARY OUTCOMES:
Objective Overall Response Rate (ORR) | From randomization to 24 month
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death. Participants needed to have two consecutive assessments of PR or CR to be a responder. Only participants with measurable disease at baseline were included in the analysis of BOR and who did not have any evaluable post-baseline assessments were classified as not evaluable.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.
Overall Survival (OS) | From randomization to 24 month
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.
  The OS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
Progression-Free Survival (PFS) | From randomization to 24 month
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
  The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No